CLINICAL TRIAL: NCT06849791
Title: Assessment of the Relative Bioavailability of ABBV-932 Formulations in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Oral ABBV-932 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M24-889
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- ABBV-932: Arm A (Experimental): Participants will receive a single dose of ABBV-932 Arm A on day 1 under fasting conditions.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm B (Experimental): Participants will receive a single dose of ABBV-932 Arm B on day 1 under fasting conditions.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm C (Experimental): Participants will receive a single dose of ABBV-932 Arm C on day 1 under fasting conditions.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm D (Experimental): Participants will receive a single dose of ABBV-932 Arm D on day 1 with a high-fat meal.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm E (Experimental): Participants will receive a single dose of ABBV-932 Arm E on day 1 with a high-fat meal.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm F (Experimental): Participants will receive a single dose of ABBV-932 Arm F on day 1 under fasting conditions.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm G (Experimental): Participants will receive a single dose of ABBV-932 Arm G on day 1 with a high-fat meal.
  Interventions: Drug: ABBV-932
- ABBV-932: Arm H (Experimental): Participants will receive a single dose of ABBV-932 Arm H on day 1 under fasting conditions.
  Interventions: Drug: ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
  Arms: ABBV-932: Arm A; ABBV-932: Arm C; ABBV-932: Arm E; ABBV-932: Arm F; ABBV-932: Arm G; ABBV-932: Arm H
Drug: ABBV-932 — Oral tablet
  Arms: ABBV-932: Arm B; ABBV-932: Arm D

SUMMARY:
This study will assess the relative bioavailability and effect of food on pharmacokinetics of ABBV-932 oral administration in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening and upon initial confinement. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-932 | Up to approximately 6 days
  Cmax of ABBV-932
Time to Cmax (Tmax) of ABBV-932 | Up to approximately 6 days
  Tmax of ABBV-932
Terminal Phase Elimination Rate Constant (Beta) of ABBV-932 | Up to approximately 6 days
  Terminal phase elimination rate constant (beta) of ABBV-932
Terminal Phase Elimination Half-Life (t1/2) of ABBV-932 | Up to approximately 6 days
  Terminal phase elimination half-life of ABBV-932
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-932 | Up to approximately 6 days
  AUCt of ABBV-932
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-932 | Up to approximately 6 days
  AUCinf of ABBV-932
Number of Participants Experiencing Adverse Events | Up to approximately 180 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 266649, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-889